CLINICAL TRIAL: NCT05539911
Title: The Effect of Using Fentanyl as an Adjuvant to Peribulbar Block to Decrease the Introaoperative Muscle Traction Pain (Proprioception) in Squint and Buckle Surgeries in Adults: RCT
Brief Title: Fentanyl as an Adjuvant to Peribulbar Block in Buckle or Squint Surgeries
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Research Institute of Ophthalmology, Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 00abeer00
Record Dates: First submitted 2022-09-10; First posted 2022-09-14 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group f (Active Comparator): patient received 50 mic fentanyl as an adjuvant to the local anesthetic mixture applied during peribulbar block in the operative eye
  Interventions: Drug: Fentanyl
- group C (Placebo Comparator): received the traditional mixture used
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Fentanyl — 50 mic fentanyl added as an adjuvant

SUMMARY:
The use of fentanyl as an adjuvant to local anesthetic mixture in many regional blocks. It was effective when used in peribulbar block in cataract and vitreoretinal surgeries.

Our study will assess its efficacy in abolishing pain during muscle traction which is usually a complain for many patients a reason to use systemic opioid intra operatively or even general anesthesia

DETAILED DESCRIPTION:
After the patient enters the OR room, an intravenous cannula will be introduced, pulse oximeter, ECG and NIBP monitors will be connected.

Nasal oxygen cannula connected; 10 ml of local anesthetic mixture is injected depending on the group the patient is allocated.

Increments of intravenous intravenous fentanyl and midazolam will be given if patient experienced unbearable pain.

All patient received peribulbar block by an experienced anesthesiologist, both patient and anesthesiologist were blinded to the drug mixture used.

Each patient received 10 ml of the anesthetic mixture according to his/ her group.

The patient was asked to fix his eyes looking straight forward toward the ceiling while lying in a supine position. A 10 ml syringe with a 25G needle was used for the local anesthetic injection. After negative aspiration, the first 5 ml were slowly injected at the junction of the lateral one third and medial two thirds of the inferior orbital margin with the bevel directed towards the equator of the eye ball parallel to the orbital floor and the other 5 ml were given between the caruncle and the medial canthus. Intermittent gentle massage was applied for 10 minutes. After satisfactory sensory and motor block, oxygen 3 L/min was delivered through a nasal cannula to the patient. Surgery was then allowed to proceed.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1, 2 & 3
* Age 18 to 70
* Patients undergoing squint or buckle surgeries

Exclusion Criteria:

* Sensitivity to any drug used in this study
* Refusal of the patient for peribulbar block
* Redo squint surgeries or previous buckle insertion
* High axial length if documented
* mentally retarded patients and
* failure of proper communication as in deafness,
* coagulation abnormalities (INR>1.4),
* infection at the injection site

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
pain during muscle traction | Intraoperative period
  numeric rating Scale for pain a scale from 0 to 10 where 0 is no pain and 10 is unbearable pain

SECONDARY OUTCOMES:
surgeon satisfaction | intraoperative
  yes or no

CONTACTS AND LOCATIONS:
Overall Officials: Abeer S Salem, MD, Principal Investigator — Research Institute of Ophthalmology
Locations (1):
- Research Institute of Ophthalmology, Giza, Egypt